CLINICAL TRIAL: NCT00139022
Title: Can Obstructive Sleep Apnea be Diagnosed at Home? A Randomised Trial of Home vs.in-Lab Diagnosis and Treatment of OSA.
Brief Title: Home Diagnosis and Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-REB# 04-91
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea, home monitoring, CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Microcephaly, Primary Autosomal Recessive, 6 | interventions — Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure

SUMMARY:
Obstructive Sleep Apnea (OSA) is a common and underrecognised condition. The diagnosis of OSA is typically made after an in-lab polysomnography (PSG) which requires an overnight stay in a sleep laboratory. Many sleep laboratories have long waiting lists for PSG. There are a number of portable devices which may be useful in home diagnosis of OSA, however there is limited data on outcomes of OSA diagnosed and treated at home. In this study we propose to compare diagnostic accuracy of a home monitoring device with a PSG and outcomes of OSA therapy when implemented at home vs in the sleep laboratory.

DETAILED DESCRIPTION:
We will randomise patients suspected to have OSA to either home evaluation and treatment (using a portable monitor and auto-CPAP) or in-lab evaluation with a PSG and manually-titrated CPAP. We will obtain sleep, sleepiness and quality of life questionnaires, vigilance testing and blood pressure at baseline and after 1, 2, 4 and 12 weeks of therapy. We will also assess and compare compliance with CPAP therapy in each arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* adult ( age > 18)
* suspected OSA
* no coexisting heart or lung disease
* not in a safety-sensitive occupation

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Sleepiness score

SECONDARY OUTCOMES:
Quality of life
Vigilance tests
Sleep quality
CPAP compliance

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Skomro, MD, Principal Investigator — Univerisity of Saskatchewan
Locations (1):
- Sleep Disorders Center, Royal Univerisity Hospital, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Skomro RP, Gjevre J, Reid J, McNab B, Ghosh S, Stiles M, Jokic R, Ward H, Cotton D. Outcomes of home-based diagnosis and treatment of obstructive sleep apnea. Chest. 2010 Aug;138(2):257-63. doi: 10.1378/chest.09-0577. Epub 2010 Feb 19. PMID 20173052